CLINICAL TRIAL: NCT05466604
Title: Comparison of the Effects of Hyaluronidase and Dexamethasone on Reduction of Postoperative Edema in Impacted Wisdom Teeth Surgery
Brief Title: Comparison of Hyaluronidase and Dexametasone in Reduction of Postoperative Edema
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Onur Koç, Doctor, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: YDU/2019//74-921
Record Dates: First submitted 2022-07-13; First posted 2022-07-20 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Edema; Pain; Trismus; Infection, Surgical Site
Keywords: postoperative edema; wisdom teeth; trismus; pain control; wound infection
MeSH Terms: conditions — Edema; Pain; Trismus; Surgical Wound Infection; Agnosia; Wound Infection

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- hyaluronidase (Experimental)
  Interventions: Drug: Hyaluronidase Injection mesomedica
- hyaluronidase control (No Intervention)
- dexamethasone (Experimental)
  Interventions: Drug: Dexamethasone dekort
- dexamethasone control (No Intervention)

INTERVENTIONS:
Drug: Hyaluronidase Injection mesomedica — injection of 150 IU hyaluronidase to perioperative region, submucosally.
  Arms: hyaluronidase
Drug: Dexamethasone dekort — injection of 8 mg dexamethasone to perioperative region, submucosally.
  Arms: dexamethasone

SUMMARY:
The present study is designed to reveal effectiveness of hyaluronidase and dexamethasone on reduction of postoperative edema, pain, trismus, and infection. For this purpose, 60 participants with symmetrical mandibular wisdom teeth enrolled the present study. All measurements and evaluations were performed before and 1, 2, 3, and 7 days later the operation.

ELIGIBILITY:
Inclusion Criteria:

* symmetrical mandibular wisdom teeth with bone retention
* patients who are signed informed consent and acceptance of study involvement forms

Exclusion Criteria:

* existence of any systemic disease
* existence of any periodical drug intake
* existence of difference in operation times of right and left impacted wisdom teeth extractions more than 5 minutes
* existence of pregnancy
* existence of breastfeeding

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
evaluation of the increase of edema in postoperative 1. day using a measuring tape in hyaluronidase experimental group | postoperative 1. day
  preoperative edema amount was subtracted from edema amount in 1. day in hyaluronidase experimental group
evaluation of the increase of edema in postoperative 2. day using a measuring tape in hyaluronidase experimental group | postoperative 2. day
  preoperative edema amount was subtracted from edema amount in 2. day in hyaluronidase experimental group
evaluation of the increase of edema in postoperative 3. day using a measuring tape in hyaluronidase experimental group | postoperative 3. day
  preoperative edema amount was subtracted from edema amount in 3. day in hyaluronidase experimental group
evaluation of the increase of edema in postoperative 7. day using a measuring tape in hyaluronidase experimental group | postoperative 7. day
  preoperative edema amount was subtracted from edema amount in 7. day in hyaluronidase experimental group
evaluation of the increase of edema in postoperative 1. day using a measuring tape in hyaluronidase control group | postoperative 1. day
  preoperative edema amount was subtracted from edema amount in 1. day in hyaluronidase control group
evaluation of the increase of edema in postoperative 2. day using a measuring tape in hyaluronidase control group | postoperative 2. day
  preoperative edema amount was subtracted from edema amount in 2. day in hyaluronidase control group
evaluation of the increase of edema in postoperative 3. day using a measuring tape in hyaluronidase control group | postoperative 3. day
  preoperative edema amount was subtracted from edema amount in 3. day in hyaluronidase control group
evaluation of the increase of edema in postoperative 7. day using a measuring tape in hyaluronidase control group | postoperative 7. day
  preoperative edema amount was subtracted from edema amount in 7. day in hyaluronidase control group
evaluation of the increase of edema in postoperative 1. day using a measuring tape in dexamethasone experimental group | postoperative 1. day
  preoperative edema amount was subtracted from edema amount in 1. day in dexamethasone experimental group
evaluation of the increase of edema in postoperative 2. day using a measuring tape in dexamethasone experimental group | postoperative 2. day
  preoperative edema amount was subtracted from edema amount in 2. day in dexamethasone experimental group
evaluation of the increase of edema in postoperative 3. day using a measuring tape in dexamethasone experimental group | postoperative 3. day
  preoperative edema amount was subtracted from edema amount in 3. day in dexamethasone experimental group
evaluation of the increase of edema in postoperative 7. day using a measuring tape in dexamethasone experimental group | postoperative 7. day
  preoperative edema amount was subtracted from edema amount in 7. day in dexamethasone experimental group
evaluation of the increase of edema in postoperative 1. day using a measuring tape in dexamethasone control group | postoperative 1. day
  preoperative edema amount was subtracted from edema amount in 1. day in dexamethasone controlgroup
evaluation of the increase of edema in postoperative 2. day using a measuring tape in dexamethasone control group | postoperative 2. day
  preoperative edema amount was subtracted from edema amount in 2. day in dexamethasone controlgroup
evaluation of the increase of edema in postoperative 3. day using a measuring tape in dexamethasone control group | postoperative 3. day
  preoperative edema amount was subtracted from edema amount in 3. day in dexamethasone controlgroup
evaluation of the increase of edema in postoperative 7. day using a measuring tape in dexamethasone control group | postoperative 7. day
  preoperative edema amount was subtracted from edema amount in 7. day in dexamethasone controlgroup
evaluation of the difference in increase amounts of edema between hyaluronidase experimental and hyaluronidase control groups in postoperative 1. day using a measuring tape | postoperative 1. day
  edema increase amount of hyaluronidase experimental group was compared with that of hyaluronidase control group in postoperative 1. day
evaluation of the difference in increase amounts of edema between hyaluronidase experimental and hyaluronidase control groups in postoperative 2. day using a measuring tape | postoperative 2. day
  edema increase amount of hyaluronidase experimental group was compared with that of hyaluronidase control group in postoperative 2. day
evaluation of the difference in increase amounts of edema between hyaluronidase experimental and hyaluronidase control groups in postoperative 3. day using a measuring tape | postoperative 3. day
  edema increase amount of hyaluronidase experimental group was compared with that of hyaluronidase control group in postoperative 3. day
evaluation of the difference in increase amounts of edema between hyaluronidase experimental and hyaluronidase control groups in postoperative 7. day using a measuring tape | postoperative 7. day
  edema increase amount of hyaluronidase experimental group was compared with that of hyaluronidase control group in postoperative 7. day
evaluation of the difference in increase amounts of edema between dexamethasone experimental and dexamethasone control groups in postoperative 1. day using a measuring tape | postoperative 1. day
  edema increase amount of dexamethasone experimental group was compared with that of dexamethasone control group in postoperative 1. day
evaluation of the difference in increase amounts of edema between dexamethasone experimental and dexamethasone control groups in postoperative 2. day using a measuring tape | postoperative 2. day
  edema increase amount of dexamethasone experimental group was compared with that of dexamethasone control group in postoperative 2. day
evaluation of the difference in increase amounts of edema between dexamethasone experimental and dexamethasone control groups in postoperative 3. day using a measuring tape | postoperative 3. day
  edema increase amount of dexamethasone experimental group was compared with that of dexamethasone control group in postoperative 3. day
evaluation of the difference in increase amounts of edema between dexamethasone experimental and dexamethasone control groups in postoperative 7. day using a measuring tape | postoperative 7. day
  edema increase amount of dexamethasone experimental group was compared with that of dexamethasone control group in postoperative 7. day
evaluation of the pain using visual analog scale (VAS) and daily count of NSAİ drug intake in hyaluronidase experimental group in postoperative 1. day | postoperative 1. day
  pain intensity of the patients in hyaluronidase experimental group was assessed using visual analog scale (VAS) and daily count of NSAİ drug intake in postoperative 1. day
evaluation of the pain using visual analog scale (VAS) and daily count of NSAİ drug intake in hyaluronidase experimental group in postoperative 2. day | postoperative 2. day
  pain intensity of the patients in hyaluronidase experimental group was assessed using visual analog scale (VAS) and daily count of NSAİ drug intake in postoperative 2. day
evaluation of the pain using visual analog scale (VAS) and daily count of NSAİ drug intake in hyaluronidase experimental group in postoperative 3. day | postoperative 3. day
  pain intensity of the patients in hyaluronidase experimental group was assessed using visual analog scale (VAS) and daily count of NSAİ drug intake in postoperative 3. day
evaluation of the pain using visual analog scale (VAS) and daily count of NSAİ drug intake in hyaluronidase experimental group in postoperative 4. day | postoperative 4. day
  pain intensity of the patients in hyaluronidase experimental group was assessed using visual analog scale (VAS) and daily count of NSAİ drug intake in postoperative 4. day
evaluation of the pain using visual analog scale (VAS) and daily count of NSAİ drug intake in hyaluronidase experimental group in postoperative 5. day | postoperative 5. day
  pain intensity of the patients in hyaluronidase experimental group was assessed using visual analog scale (VAS) and daily count of NSAİ drug intake in postoperative 5. day
evaluation of the pain using visual analog scale (VAS) and daily count of NSAİ drug intake in hyaluronidase experimental group in postoperative 6. day | postoperative 6. day
  pain intensity of the patients in hyaluronidase experimental group was assessed using visual analog scale (VAS) and daily count of NSAİ drug intake in postoperative 6. day
evaluation of the pain using visual analog scale (VAS) and daily count of NSAİ drug intake in hyaluronidase experimental group in postoperative 7. day | postoperative 7. day
  pain intensity of the patients in hyaluronidase experimental group was assessed using visual analog scale (VAS) and daily count of NSAİ drug intake in postoperative 7. day
evaluation of the pain using visual analog scale (VAS) and daily count of NSAİ drug intake in hyaluronidase control group in postoperative 1. day | postoperative 1. day
  pain intensity of the patients in hyaluronidase control group was assessed using visual analog scale (VAS) and daily count of NSAİ drug intake in postoperative 1. day
evaluation of the pain using visual analog scale (VAS) and daily count of NSAİ drug intake in hyaluronidase control group in postoperative 2. day | postoperative 2. day
  pain intensity of the patients in hyaluronidase control group was assessed using visual analog scale (VAS) and daily count of NSAİ drug intake in postoperative 2. day
evaluation of the pain using visual analog scale (VAS) and daily count of NSAİ drug intake in hyaluronidase control group in postoperative 3. day | postoperative 3. day
  pain intensity of the patients in hyaluronidase control group was assessed using visual analog scale (VAS) and daily count of NSAİ drug intake in postoperative 3. day
evaluation of the pain using visual analog scale (VAS) and daily count of NSAİ drug intake in hyaluronidase control group in postoperative 4. day | postoperative 4. day
  pain intensity of the patients in hyaluronidase control group was assessed using visual analog scale (VAS) and daily count of NSAİ drug intake in postoperative 4. day
evaluation of the pain using visual analog scale (VAS) and daily count of NSAİ drug intake in hyaluronidase control group in postoperative 5. day | postoperative 5. day
  pain intensity of the patients in hyaluronidase control group was assessed using visual analog scale (VAS) and daily count of NSAİ drug intake in postoperative 5. day
evaluation of the pain using visual analog scale (VAS) and daily count of NSAİ drug intake in hyaluronidase control group in postoperative 6. day | postoperative 6. day
  pain intensity of the patients in hyaluronidase control group was assessed using visual analog scale (VAS) and daily count of NSAİ drug intake in postoperative 6. day
evaluation of the pain using visual analog scale (VAS) and daily count of NSAİ drug intake in hyaluronidase control group in postoperative 7. day | postoperative 7. day
  pain intensity of the patients in hyaluronidase control group was assessed using visual analog scale (VAS) and daily count of NSAİ drug intake in postoperative 7. day
evaluation of the pain using visual analog scale (VAS) and daily count of NSAİ drug intake in dexamethasone experimental group in postoperative 1. day | postoperative 1. day
  pain intensity of the patients in dexamethasone experimental group was assessed using visual analog scale (VAS) and daily count of NSAİ drug intake in postoperative 1. day
evaluation of the pain using visual analog scale (VAS) and daily count of NSAİ drug intake in dexamethasone experimental group in postoperative 2. day | postoperative 2. day
  pain intensity of the patients in dexamethasone experimental group was assessed using visual analog scale (VAS) and daily count of NSAİ drug intake in postoperative 2. day
evaluation of the pain using visual analog scale (VAS) and daily count of NSAİ drug intake in dexamethasone experimental group in postoperative 3. day | postoperative 3. day
  pain intensity of the patients in dexamethasone experimental group was assessed using visual analog scale (VAS) and daily count of NSAİ drug intake in postoperative 3. day
evaluation of the pain using visual analog scale (VAS) and daily count of NSAİ drug intake in dexamethasone experimental group in postoperative 4. day | postoperative 4. day
  pain intensity of the patients in dexamethasone experimental group was assessed using visual analog scale (VAS) and daily count of NSAİ drug intake in postoperative 4. day
evaluation of the pain using visual analog scale (VAS) and daily count of NSAİ drug intake in dexamethasone experimental group in postoperative 5. day | postoperative 5. day
  pain intensity of the patients in dexamethasone experimental group was assessed using visual analog scale (VAS) and daily count of NSAİ drug intake in postoperative 5. day
evaluation of the pain using visual analog scale (VAS) and daily count of NSAİ drug intake in dexamethasone experimental group in postoperative 6. day | postoperative 6. day
  pain intensity of the patients in dexamethasone experimental group was assessed using visual analog scale (VAS) and daily count of NSAİ drug intake in postoperative 6. day
evaluation of the pain using visual analog scale (VAS) and daily count of NSAİ drug intake in dexamethasone experimental group in postoperative 7. day | postoperative 7. day
  pain intensity of the patients in dexamethasone experimental group was assessed using visual analog scale (VAS) and daily count of NSAİ drug intake in postoperative 7. day
evaluation of the pain using visual analog scale (VAS) and daily count of NSAİ drug intake in dexamethasone control group in postoperative 1. day | postoperative 1. day
  pain intensity of the patients in dexamethasone control group was assessed using visual analog scale (VAS) and daily count of NSAİ drug intake in postoperative 1. day
evaluation of the pain using visual analog scale (VAS) and daily count of NSAİ drug intake in dexamethasone control group in postoperative 2. day | postoperative 2. day
  pain intensity of the patients in dexamethasone control group was assessed using visual analog scale (VAS) and daily count of NSAİ drug intake in postoperative 2. day
evaluation of the pain using visual analog scale (VAS) and daily count of NSAİ drug intake in dexamethasone control group in postoperative 3. day | postoperative 3. day
  pain intensity of the patients in dexamethasone control group was assessed using visual analog scale (VAS) and daily count of NSAİ drug intake in postoperative 3. day
evaluation of the pain using visual analog scale (VAS) and daily count of NSAİ drug intake in dexamethasone control group in postoperative 4. day | postoperative 4. day
  pain intensity of the patients in dexamethasone control group was assessed using visual analog scale (VAS) and daily count of NSAİ drug intake in postoperative 4. day
evaluation of the pain using visual analog scale (VAS) and daily count of NSAİ drug intake in dexamethasone control group in postoperative 5. day | postoperative 5. day
  pain intensity of the patients in dexamethasone control group was assessed using visual analog scale (VAS) and daily count of NSAİ drug intake in postoperative 5. day
evaluation of the pain using visual analog scale (VAS) and daily count of NSAİ drug intake in dexamethasone control group in postoperative 6. day | postoperative 6. day
  pain intensity of the patients in dexamethasone control group was assessed using visual analog scale (VAS) and daily count of NSAİ drug intake in postoperative 6. day
evaluation of the pain using visual analog scale (VAS) and daily count of NSAİ drug intake in dexamethasone control group in postoperative 7. day | postoperative 7. day
  pain intensity of the patients in dexamethasone control group was assessed using visual analog scale (VAS) and daily count of NSAİ drug intake in postoperative 7. day
evaluation of trismus using a ruler, which measures the opening between mandibular and maxillary right first incisors of hyaluronidase experimental group preoperatively. | preoperative
  amount of trismus is revealed measuring the distance between the tips of incisal edges of mandibular and maxillary right first incisors using a ruler
evaluation of trismus using a ruler, which measures the opening between mandibular and maxillary right first incisors of hyaluronidase experimental group in postoperative 1. day. | postoperative 1. day
  amount of trismus is revealed measuring the distance between the tips of incisal edges of mandibular and maxillary right first incisors using a ruler
evaluation of trismus using a ruler, which measures the opening between mandibular and maxillary right first incisors of hyaluronidase experimental group in postoperative 2. day. | postoperative 2. day
  amount of trismus is revealed measuring the distance between the tips of incisal edges of mandibular and maxillary right first incisors using a ruler
evaluation of trismus using a ruler, which measures the opening between mandibular and maxillary right first incisors of hyaluronidase experimental group in postoperative 3. day. | postoperative 3. day
  amount of trismus is revealed measuring the distance between the tips of incisal edges of mandibular and maxillary right first incisors using a ruler
evaluation of trismus using a ruler, which measures the opening between mandibular and maxillary right first incisors of hyaluronidase experimental group in postoperative 7. day. | postoperative 7. day
  amount of trismus is revealed measuring the distance between the tips of incisal edges of mandibular and maxillary right first incisors using a ruler
evaluation of trismus using a ruler, which measures the opening between mandibular and maxillary right first incisors of hyaluronidase control group preoperatively. | preoperative
  amount of trismus is revealed measuring the distance between the tips of incisal edges of mandibular and maxillary right first incisors using a ruler
evaluation of trismus using a ruler, which measures the opening between mandibular and maxillary right first incisors of hyaluronidase control group in postoperative 1. day. | postoperative 1. day
  amount of trismus is revealed measuring the distance between the tips of incisal edges of mandibular and maxillary right first incisors using a ruler
evaluation of trismus using a ruler, which measures the opening between mandibular and maxillary right first incisors of hyaluronidase control group in postoperative 2. day. | postoperative 2. day
  amount of trismus is revealed measuring the distance between the tips of incisal edges of mandibular and maxillary right first incisors using a ruler
evaluation of trismus using a ruler, which measures the opening between mandibular and maxillary right first incisors of hyaluronidase control group in postoperative 3. day. | postoperative 3. day
  amount of trismus is revealed measuring the distance between the tips of incisal edges of mandibular and maxillary right first incisors using a ruler
evaluation of trismus using a ruler, which measures the opening between mandibular and maxillary right first incisors of hyaluronidase control group in postoperative 7. day. | postoperative 7. day
  amount of trismus is revealed measuring the distance between the tips of incisal edges of mandibular and maxillary right first incisors using a ruler
evaluation of trismus using a ruler, which measures the opening between mandibular and maxillary right first incisors of dexamethasone experimental group preoperatively. | preoperative
  amount of trismus is revealed measuring the distance between the tips of incisal edges of mandibular and maxillary right first incisors using a ruler
evaluation of trismus using a ruler, which measures the opening between mandibular and maxillary right first incisors of dexamethasone experimental group in postoperative 1. day. | postoperative 1. day
  amount of trismus is revealed measuring the distance between the tips of incisal edges of mandibular and maxillary right first incisors using a ruler
evaluation of trismus using a ruler, which measures the opening between mandibular and maxillary right first incisors of dexamethasone experimental group in postoperative 2. day. | postoperative 2. day
  amount of trismus is revealed measuring the distance between the tips of incisal edges of mandibular and maxillary right first incisors using a ruler
evaluation of trismus using a ruler, which measures the opening between mandibular and maxillary right first incisors of dexamethasone experimental group in postoperative 3. day. | postoperative 3. day
  amount of trismus is revealed measuring the distance between the tips of incisal edges of mandibular and maxillary right first incisors using a ruler
evaluation of trismus using a ruler, which measures the opening between mandibular and maxillary right first incisors of dexamethasone experimental group in postoperative 7. day. | postoperative 7. day
  amount of trismus is revealed measuring the distance between the tips of incisal edges of mandibular and maxillary right first incisors using a ruler
evaluation of trismus using a ruler, which measures the opening between mandibular and maxillary right first incisors of dexamethasone control group preoperatively. | preoperative
  amount of trismus is revealed measuring the distance between the tips of incisal edges of mandibular and maxillary right first incisors using a ruler
evaluation of trismus using a ruler, which measures the opening between mandibular and maxillary right first incisors of dexamethasone control group in postoperative 1. day. | postoperative 1. day
  amount of trismus is revealed measuring the distance between the tips of incisal edges of mandibular and maxillary right first incisors using a ruler
evaluation of trismus using a ruler, which measures the opening between mandibular and maxillary right first incisors of dexamethasone control group in postoperative 2. day. | postoperative 2. day
  amount of trismus is revealed measuring the distance between the tips of incisal edges of mandibular and maxillary right first incisors using a ruler
evaluation of trismus using a ruler, which measures the opening between mandibular and maxillary right first incisors of dexamethasone control group in postoperative 3. day. | postoperative 3. day
  amount of trismus is revealed measuring the distance between the tips of incisal edges of mandibular and maxillary right first incisors using a ruler
evaluation of trismus using a ruler, which measures the opening between mandibular and maxillary right first incisors of dexamethasone control group in postoperative 7. day. | postoperative 7. day
  amount of trismus is revealed measuring the distance between the tips of incisal edges of mandibular and maxillary right first incisors using a ruler
evaluation of infection in operation site via determination of infection signs in physical examination of hyaluronidase experimental group preoperatively. | preoperative
  existence of infection signs were determined using physical examination method. if the count of + signs are more than half of total amount of determined signs, the evaluation is accepted as (+) infected.
evaluation of infection in operation site via determination of infection signs in physical examination of hyaluronidase experimental group in postoperative 1. day. | postoperative 1. day
  existence of infection signs were determined using physical examination method. if the count of + signs are more than half of total amount of determined signs, the evaluation is accepted as (+) infected.
evaluation of infection in operation site via determination of infection signs in physical examination of hyaluronidase experimental group in postoperative 2. day. | postoperative 2. day
  existence of infection signs were determined using physical examination method. if the count of + signs are more than half of total amount of determined signs, the evaluation is accepted as (+) infected.
evaluation of infection in operation site via determination of infection signs in physical examination of hyaluronidase experimental group in postoperative 3. day. | postoperative 3. day
  existence of infection signs were determined using physical examination method. if the count of + signs are more than half of total amount of determined signs, the evaluation is accepted as (+) infected.
evaluation of infection in operation site via determination of infection signs in physical examination of hyaluronidase experimental group in postoperative 7. day. | postoperative 7. day
  existence of infection signs were determined using physical examination method. if the count of + signs are more than half of total amount of determined signs, the evaluation is accepted as (+) infected.
evaluation of infection in operation site via determination of infection signs in physical examination of hyaluronidase control group preoperatively. | preoperative
  existence of infection signs were determined using physical examination method. if the count of + signs are more than half of total amount of determined signs, the evaluation is accepted as (+) infected.
evaluation of infection in operation site via determination of infection signs in physical examination of hyaluronidase control group in postoperative 1. day. | postoperative 1. day
  existence of infection signs were determined using physical examination method. if the count of + signs are more than half of total amount of determined signs, the evaluation is accepted as (+) infected.
evaluation of infection in operation site via determination of infection signs in physical examination of hyaluronidase control group in postoperative 2. day. | postoperative 2. day
  existence of infection signs were determined using physical examination method. if the count of + signs are more than half of total amount of determined signs, the evaluation is accepted as (+) infected.
evaluation of infection in operation site via determination of infection signs in physical examination of hyaluronidase control group in postoperative 3. day. | postoperative 3. day
  existence of infection signs were determined using physical examination method. if the count of + signs are more than half of total amount of determined signs, the evaluation is accepted as (+) infected.
evaluation of infection in operation site via determination of infection signs in physical examination of hyaluronidase control group in postoperative 7. day. | postoperative 7. day
  existence of infection signs were determined using physical examination method. if the count of + signs are more than half of total amount of determined signs, the evaluation is accepted as (+) infected.
evaluation of infection in operation site via determination of infection signs in physical examination of dexamethasone experimental group preoperatively. | preoperative
  existence of infection signs were determined using physical examination method. if the count of + signs are more than half of total amount of determined signs, the evaluation is accepted as (+) infected.
evaluation of infection in operation site via determination of infection signs in physical examination of dexamethasone experimental group in postoperative 1. day | postoperative 1. day
  existence of infection signs were determined using physical examination method. if the count of + signs are more than half of total amount of determined signs, the evaluation is accepted as (+) infected.
evaluation of infection in operation site via determination of infection signs in physical examination of dexamethasone experimental group in postoperative 2. day | postoperative 2. day
  existence of infection signs were determined using physical examination method. if the count of + signs are more than half of total amount of determined signs, the evaluation is accepted as (+) infected.
evaluation of infection in operation site via determination of infection signs in physical examination of dexamethasone experimental group in postoperative 3. day | postoperative 3. day
  existence of infection signs were determined using physical examination method. if the count of + signs are more than half of total amount of determined signs, the evaluation is accepted as (+) infected.
evaluation of infection in operation site via determination of infection signs in physical examination of dexamethasone experimental group in postoperative 7. day | postoperative 7. day
  existence of infection signs were determined using physical examination method. if the count of + signs are more than half of total amount of determined signs, the evaluation is accepted as (+) infected.
evaluation of infection in operation site via determination of infection signs in physical examination of dexamethasone control group preoperatively. | preoperatively
  existence of infection signs were determined using physical examination method. if the count of + signs are more than half of total amount of determined signs, the evaluation is accepted as (+) infected.
evaluation of infection in operation site via determination of infection signs in physical examination of dexamethasone control group in postoperative 1. day | postoperative 1. day
  existence of infection signs were determined using physical examination method. if the count of + signs are more than half of total amount of determined signs, the evaluation is accepted as (+) infected.
evaluation of infection in operation site via determination of infection signs in physical examination of dexamethasone control group in postoperative 2. day | postoperative 2. day
  existence of infection signs were determined using physical examination method. if the count of + signs are more than half of total amount of determined signs, the evaluation is accepted as (+) infected.
evaluation of infection in operation site via determination of infection signs in physical examination of dexamethasone control group in postoperative 3. day | postoperative 3. day
  existence of infection signs were determined using physical examination method. if the count of + signs are more than half of total amount of determined signs, the evaluation is accepted as (+) infected.
evaluation of infection in operation site via determination of infection signs in physical examination of dexamethasone control group in postoperative 7. day | postoperative 7. day
  existence of infection signs were determined using physical examination method. if the count of + signs are more than half of total amount of determined signs, the evaluation is accepted as (+) infected.

CONTACTS AND LOCATIONS:
Locations (2):
- Near East University, Nicosia, Cyprus
- Hacettepe University, Ankara, Sıhhiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Koc O, Er N, Karaca C, Bilginaylar K. Comparison of the effects of submucosal hyaluronidase and dexamethasone on postoperative edema, pain, trismus, and infection following impacted third molar surgery. BMC Oral Health. 2024 Aug 30;24(1):1018. doi: 10.1186/s12903-024-04729-1. PMID 39215323